CLINICAL TRIAL: NCT06488924
Title: An Open-label Phase I/II Study of JR-446 in Mucopolysaccharidosis Type IIIB
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-446-101
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis III-B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JR-446 (Experimental)
  Interventions: Drug: JR-446

INTERVENTIONS:
Drug: JR-446 — IV infusion

SUMMARY:
A Phase I/ II, open-label study, designed to evaluate the safety and explore efficacy of the study drug in development for the treatment of MPS IIIB patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age of <18 years
* Confirmed diagnosis of MPS IIIB

Exclusion Criteria:

* Prior experience to gene therapy or HSCT with successful engraftment
* Past use of another investigational drug or product in last 4 months or 5 half-lives (whichever is longer) before signing ICF
* Current participation in a clinical trial or past participation (within 30 days of enrolment into this study) in a study involving invasive procedures
* Past use of Genistein or Kineret (anakinra) within 4 months before signing ICF
* Serious drug allergy or hypersensitivity
* Contraindication for lumbar puncture or MRI
* History of bleeding disorder or current use of medications that, in the opinion of the investigator, place them at risk of bleeding following lumbar puncture

The above information is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
To establish the safety and tolerability of JR-446 in MPSIIIB patients | up to 4 years (multiple visits)
To determine the pharmacodynamic effects of JR-446 in MPSIIIB patients | up to 4 years (multiple visits)

SECONDARY OUTCOMES:
To assess PK profile of JR-446 in MPSIIIB patients | up to 4 years (multiple visits)
To explore the potential efficacy of JR-446 in the treatment of patients with MPS IIIB | up to 4 years (multiple visits)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Hiroshima University Hospital, Hiroshima
  - University of the Ryukyus Hospital, Okinawa
  - National Center for Child Health and Development, Tokyo